CLINICAL TRIAL: NCT01841164
Title: A Study of the Effects of the Selective CysLT1 Antagonist Montelukast on Bronchoconstriction and Airway Inflammation Induced by Inhalation of Leukotriene E4 in Subjects With Asthma
Brief Title: A Mechanistic Study to Evaluate the Efficacy of Montelukast on Airway Function in Asthma
Acronym: E-Type
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Barbro Dahlen, Senior Consultant, MD PhD, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E-Type 4 KI_Cfa
Record Dates: First submitted 2013-04-15; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
Keywords: Leukotriene responsiveness; LTE4; asthma; airway hyperresponsiveness; bronchoprovocation; anti-asthmatic agents; human
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — montelukast; Leukotriene E4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Experimental): 5 to 7 days of treatment with montelukast 10 mg 2 tablets bid. Efficacy of treatment is evaluated on airway responsiveness to inhaled leukotriene E4.
  Interventions: Drug: Montelukast; Other: Inhaled leukotriene E4
- Sugar pill (Placebo Comparator): Placebo for montelukast 5-7 days 2 tablets bid. Efficacy of treatment is evaluated on airway responsiveness to inhaled leukotriene E4.
  Interventions: Drug: Placebo for montelukast; Other: Inhaled leukotriene E4

INTERVENTIONS:
Drug: Montelukast
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo for montelukast — Sugar pills manufactured to mimic Singulair
  Arms: Sugar pill
Other: Inhaled leukotriene E4 — Inhalation challenge with aerosolized GMP-grade LTE4 (Cayman Chemical Company 1180 East Ellsworth Road, Ann Arbor, Michigan 48108,USA)
  Other Names: LTE4

SUMMARY:
The trial is an investigator-driven research study in subjects with intermittent asthma, the aim of which is to explore the likelihood of a functionally important separate leukotriene E4 (LTE4) receptor in airways and/or inflammatory cells in human subjects with asthma.

Mostly on the basis of experiments in mice models, the prevailing view suggests that the present class of anti-leukotriene drugs are insufficient because they do not block the pro-inflammatory and bronchoconstrictive effects of LTE4. It is established by us and other groups that LTE4 is the most stable and long-lived leukotriene.

The study will establish the effect of oral treatment with the highly selective CysLT1-receptor antagonist, montelukast, on bronchial responsiveness to inhaled LTE4 in subjects with intermittent asthma

DETAILED DESCRIPTION:
Rationale: It has been proposed that there is a specific LTE4-receptor which causes infiltration of inflammatory cells and bronchoconstriction. This receptor is not blocked by the current class of clinically used antileukotriene drugs. The proposal receives circumstantial support from animal models, but has not been tested in a controlled study in subjects with asthma.

Study design: The study will have a placebo-controlled, double-blind, randomised, cross-over design. A screening period will precede the randomized phase. This will include routine haematology, blood chemistry and urinalyses, baseline measurements of exhaled nitric oxide, airway responsiveness to inhaled methacholine and, on a separate day, airway responsiveness to inhaled LTE4. Provided the subjects fulfill inclusion but not exclusion criteria, subjects will be randomized to receive medication with montelukast or matching placebo for 5 to 7 days. The intervention will be evaluated in the inhalation challenge setting using a rising dose cumulative protocol for inhaled LTE4 to induce a standardised bronchoconstriction (25% drop in lung function). The LTE4 challenge test is performed on the last treatment day, with the last dose of study medication taken in the research laboratory. Sampling of urine, blood and induced sputum will be done for measurements of lipid mediators and cellular responses.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18-55 years inclusive
2. Have a diagnosed history of asthma as defined by at least one of the following:

   1. response to standard asthma treatment
   2. episodic wheezing
   3. change in lung function over short periods of time
3. Be a non-smoker for the last two years and a total of smoking less than 5 pack-years
4. Display a positive methacholine challenge test as evidenced by a PD20 (provocative dose causing 20% fall in forced expiratory volume in one second) ≤ 3621 µg cumulated dose within 8 weeks prior to screening or at the screening visit.
5. Have stable intermittent asthma, only using bronchodilator therapy as needed for the last 4 weeks.
6. Produce FEV1 (forced expiratory volume in one second) ≥ 70 % of predicted

   -

Exclusion Criteria:

1. Any significant respiratory disease, other than asthma.
2. Subjects with seasonal asthma may not be included if they are in their season.
3. Use of:

   * oral or inhaled glucocorticosteroid treatment for the last 4 weeks prior to inclusion or during the study
   * inhaled long-acting or oral beta2-agonists, anticholinergic bronchodilators, antihistamines, theophyllines, chromones and antileukotrienes within 2 weeks of screening
   * regular NSAIDs
   * drugs that inhibit the enzyme CYP3A (e.g. ritonavir, azol, antifungals, macrolides)
   * beta-blocking agents
4. Upper or lower respiratory tract infection within 4 weeks before inclusion
5. Evidence (from medical history or physical examination) of any disease that in the investigators mind would affect the results of the study, in particular liver disease and/or signs of liver function impairment
6. Participating in another study in the four weeks prior to screening
7. Females who are pregnant, intend to be or who are lactating
8. Subjects with history of aspirin-sensitive respiratory disease

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Bronchoconstriction measured as LTE4 PD20. | Up to three years
  To establish the effect of oral treatment with the highly selective CysLT1-receptor antagonist montelukast on bronchial responsiveness to inhaled LTE4 in subjects with intermittent asthma.

SECONDARY OUTCOMES:
Airway inflammation measured as sputum eosinophils | Up to three years
  To establish the effect of oral treatment with the highly selective CysLT1-receptor antagonist montelukast on airway inflammation, assessed as sputum cells, induced by inhaled LTE4, in subjects with intermittent asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Barbro Dahlen, MD PhD, Principal Investigator — Karolinska Institutet and Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Lazarinis N, Bood J, Gomez C, Kolmert J, Lantz AS, Gyllfors P, Davis A, Wheelock CE, Dahlen SE, Dahlen B. Leukotriene E4 induces airflow obstruction and mast cell activation through the cysteinyl leukotriene type 1 receptor. J Allergy Clin Immunol. 2018 Oct;142(4):1080-1089. doi: 10.1016/j.jaci.2018.02.024. Epub 2018 Mar 5. PMID 29518425